CLINICAL TRIAL: NCT05941884
Title: Possible Diagnostic Protein Markers in Schistosoma Related Bladder Diseases.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Samah Mohammad Hussein, Assistant Lecturer at Parasitology department, Assiut University
Other Study IDs: PDPMSRBD
Record Dates: First submitted 2023-06-19; First posted 2023-07-12 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Schistosoma Haematobium
MeSH Terms: conditions — Schistosomiasis haematobia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Urine sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Schistosoma haematobium cystitis.: patient has symptoms suggestive of Schistosoma haematobium infection like terminal hematuria and burning micturition
  Interventions: Diagnostic Test: microscopic examination of urine
- Healthy personnel.: as control group
  Interventions: Diagnostic Test: microscopic examination of urine
- Schistosomal bladder cancer.: from patient undergone diagnostic cystoscopy and sampling and confirmed pathologically as Schistosomal bladder cancer.
  Interventions: Diagnostic Test: Immunohistochemistry staining,; Diagnostic Test: microscopic examination of urine
- non Schistosomal bladder cancer.: from patient undergone diagnostic cystoscopy and sampling and confirmed pathologically as non Schistosomal bladder cancer.
  Interventions: Diagnostic Test: Immunohistochemistry staining,
- Schistosomal cystitis patients.: from patient undergone diagnostic cystoscopy and sampling and confirmed pathologically as Schistosomal cystitis
  Interventions: Diagnostic Test: Immunohistochemistry staining,
- healthy bladder tissue from tissue biopsy patient with benign prostatic hyperplasia.: as control group
  Interventions: Diagnostic Test: Immunohistochemistry staining,

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry staining, — Tissue samples:
  * Histopathological examination: Hematoxylin and Eosin slides will be prepared and examined.
    * The only dependable criterion for the diagnosis of bilharzial infestation is the microscopic detection of Bilharzia ova in pathological sections.
    * Pathology (cystitis- cancer and its grade staging will be reported in accordance with the 2022 World Health Organization Classification of Tumors of the Urinary System (17).
  * To quantify levels of Nuclear factor kappa B and protein kinase c α:
    * Immunohistochemistry according to the manufacturer's instructions.
  Groups: Schistosomal bladder cancer.; Schistosomal cystitis patients.; healthy bladder tissue from tissue biopsy patient with benign prostatic hyperplasia.; non Schistosomal bladder cancer.
Diagnostic Test: microscopic examination of urine — Urine samples:
  * Mic roscopic examination (detection of S. haematobium egg - egg counting)
  * Detection of HSP 70 Measurements: indirect ELISA will be used to quantify HSP concentrations in urine.
  Groups: Healthy personnel.; Schistosoma haematobium cystitis.; Schistosomal bladder cancer.

SUMMARY:
Schistosomiasis is the second most common parasitic infection affecting humans, endemic in the Middle East, especially Egypt (1), and in 42 African countries (2).

There are 5 main species infecting humans: S. mansoni, S. haematobium, S. japonicum, S. intercalatum, and S. mekongi. S. haematobium is responsible for chronic urogenital infections that may cause serious complications (3). Urinary schistosomiasis is mostly borne in rural and agricultural communities, according to WHO (4)

DETAILED DESCRIPTION:
Bleeding, anemia and chronic renal failure are common presentation. Bladder cancer is associated with schistosomiasis, However the mechanism by which it occurs is still controversial. Chronic interaction with the host immune system as well as association with other carcinogenic agents can lead to the neoplastic transformation (3). The International Agency for Research on Cancer classifies the infection with S. haematobium as a group 1 carcinogen, a definitive cause of cancer (5).

Bladder cancer (BC) is the sixth most prevalent cancer in both genders worldwide. Amongst Egyptian males, bladder cancer is the most common malignancy accounting for 16% with more than 7,900 deaths per year. The main risk factor was urinary schistosomiasis which is more frequent in Upper Egypt (1).

Urothelial carcinoma represents the most common histologic type of BC, accounting for 90% of all cases. Squamous cell carcinoma may develop following bilharziasis infection, in addition other types includes adenocarcinoma and small cell carcinoma were reported (6). The WHO classification includes urothelial papilla, papillary urothelial neoplasm of low malignant potential (PUNLMP), low-grade urothelial carcinoma (LGPUC) and high- grade UC (HGPUC) (7).

Urine cytology is the only established noninvasive adjunct to cystoscopy. Being in close contact with tumor cells and adjacent inflamed urothelium. Thus, immune mediators in urine may serve as biomarkers (8). Urine biomarkers of schistosomal bladder cancer can be used as diagnostic markers in patients, and prognostic indicators of disease survival, and as early detectors of recurrent disease in the monitored patient (9).

Heat shock proteins (HSPs) are synthesized by cells in response to various stress conditions, including carcinogenesis. These molecules have been studied in several malignancies, they may be useful markers for patients with schistosomiasis-associated bladder cancer and may be used for predicting disease progression. (10). HSPs are upregulated when cells are exposed to elevated temperature. In neoplasia, the expression of HSPs is implicated in the regulation of apoptosis and tumor-cell growth, helps tumor to evade immune surveillance. As it has been reported to abort Th1 effector immunity and enhance Th2 down- regulatory immune responses. Thus, downregulate antitumor effector T cells (8). Urine proteome profile provide deeper insights into urogenital schistosomiasis, it's carcinogenesis and highlight potential biomarkers for diagnosis and/or prognosis (11).

Immunohistochemistry (IHC) is currently the most widely used pathological technique for accurate diagnosis of urinary bladder neoplasms. Moreover, identification and validation of the prognostic IHC signature have been reported in various cancer types and proved to be a promising complement in therapeutic planning and patient management (12). As oxidative stress and immune defense systems responsible for microbicide activity are the most representative clusters in urogenital schistosomiasis patients. Proteins involved in immunity, negative regulation of endopeptidase activity, and inflammation were more prevalent in UGS patients with bladder cancer (11).

NF-ƙB was first identified in active B cells by its binding affinity to immunoglobulin enhancer. NF-ƙB serves as dominant modulator of immuno-inflammatory responses. (13). It plays a critical role in normal physiology and bladder cancer progression. NF-ƙB orchestrates protein interactions (PTEN, survivin, VEGF), regulation (CYLD, USP13) and gene expression (Trp 53) resulting in bladder cancer progression, recurrence, and resistance to therapy. Bladder cancer patients have constitutively active NF-ƙB triggered by pro-inflammatory cytokines, chemokines, and hypoxia, augmenting carcinogenesis and progression (14).

Further, Protein kinase C α (PKC) is one of the serine/threonine kinases that regulates a variety of cellular biological process, such as apoptosis. It has been firmly established that PKCs are closely related to process of tumorigenesis, including the initiation and progression of bladder cancer (15). In addition, activated PKC α is involved in bladder cancer cell proliferation, survival, invasion, migration, and anticancer drug resistance (16).

In literature, the evaluation of schistosomal infestation is not precise as it depends on the histopathologic findings, which proved to be less accurate. Most of them focused on the prognostic role of biomarkers rather than their role in diagnosis and pathogenesis.

Our aim in this study is to identify the potential causal relationship between schistosomal infection and levels of NF-kappa-B and Protein kinase C α signaling and bladder cancer development and highlights their role in bladder cancer pathogenesis

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of different age groups known to suffer from cystitis and bladder cancer regardless results from schistosomal infection or any other causes.

Exclusion Criteria:

* patients with concomitant other tumours.
* patients with other urinary tract infection.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female patients of different age groups known to suffer from cystitis and bladder cancer regardless results from schistosomal infection or any other causes.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
NF-kappa-B and Protein kinase Cα | 2 years
  Association and changes of NF-kappa-B and Protein kinase Cα as diagnostic markers in chronic schistosomaiasis with or without bladder cancer
heat shock protein | 1 year
  Changes of heat shock protein HSP 70 as urinary biomarkers for Schistosomal bladder diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma G Sayed, prof, Study Director — unaffiliation
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Amin HAA, Kobaisi MH, Samir RM. Schistosomiasis and Bladder Cancer in Egypt: Truths and Myths. Open Access Maced J Med Sci. 2019 Dec 10;7(23):4023-4029. doi: 10.3889/oamjms.2019.857. eCollection 2019 Dec 15. PMID 32165946
- [Background] Efared B, Bako ABA, Idrissa B, Alhousseini D, Boureima HS, Sode HC, Nouhou H. Urinary bladder Schistosoma haematobium-related squamous cell carcinoma: a report of two fatal cases and literature review. Trop Dis Travel Med Vaccines. 2022 Feb 15;8(1):3. doi: 10.1186/s40794-022-00161-x. PMID 35164874
- [Background] Nacif-Pimenta R, da Silva Orfano A, Mosley IA, Karinshak SE, Ishida K, Mann VH, Coelho PMZ, da Costa JMC, Hsieh MH, Brindley PJ, Rinaldi G. Differential responses of epithelial cells from urinary and biliary tract to eggs of Schistosoma haematobium and S. mansoni. Sci Rep. 2019 Jul 24;9(1):10731. doi: 10.1038/s41598-019-46917-y. PMID 31341177
- [Background] Al-Delaimy WK, Awadalla A, El-Assmy A, Abol-Enein H, Shokeir A. Comparison of urinary telomerase, CD44, and NMP22 assays for detection of bladder squamous cell carcinoma. Curr Urol. 2022 Sep;16(3):154-159. doi: 10.1097/CU9.0000000000000098. Epub 2022 Aug 2. PMID 36204357
- [Background] Chen Z, Ding W, Xu K, Tan J, Sun C, Gou Y, Tong S, Xia G, Fang Z, Ding Q. The 1973 WHO Classification is more suitable than the 2004 WHO Classification for predicting prognosis in non-muscle-invasive bladder cancer. PLoS One. 2012;7(10):e47199. doi: 10.1371/journal.pone.0047199. Epub 2012 Oct 17. PMID 23082147
- [Background] Eissa S, Matboli M, Shawky S, Essawy NO. Urine biomarkers of schistosomiais and its associated bladder cancer. Expert Rev Anti Infect Ther. 2015 Aug;13(8):985-93. doi: 10.1586/14787210.2015.1051032. Epub 2015 Jun 23. PMID 26105083
- [Background] El-Meghawry El-Kenawy A, El-Kott AF, Hasan MS. Heat shock protein expression independently predicts survival outcome in schistosomiasis-associated urinary bladder cancer. Int J Biol Markers. 2008 Oct-Dec;23(4):214-8. doi: 10.1177/172460080802300403. PMID 19199268
- [Background] Wu J, Wen JM, Wang YC, Luo WJ, Wang QF, Lv H, Dai B, Ye DW, Su HC, Zhu YP. Prognostic Value of an Immunohistochemical Signature in Patients With Bladder Cancer Undergoing Radical Cystectomy. Front Oncol. 2021 Mar 25;11:641385. doi: 10.3389/fonc.2021.641385. eCollection 2021. PMID 33842349
- [Background] Zheng J, Kong C, Yang X, Cui X, Lin X, Zhang Z. Protein kinase C-alpha (PKCalpha) modulates cell apoptosis by stimulating nuclear translocation of NF-kappa-B p65 in urothelial cell carcinoma of the bladder. BMC Cancer. 2017 Jun 19;17(1):432. doi: 10.1186/s12885-017-3401-7. PMID 28629334
- [Background] Kawano T, Tachibana Y, Inokuchi J, Kang JH, Murata M, Eto M. Identification of Activated Protein Kinase Calpha (PKCalpha) in the Urine of Orthotopic Bladder Cancer Xenograft Model as a Potential Biomarker for the Diagnosis of Bladder Cancer. Int J Mol Sci. 2021 Aug 27;22(17):9276. doi: 10.3390/ijms22179276. PMID 34502182
- [Background] Netto GJ, Amin MB, Berney DM, Comperat EM, Gill AJ, Hartmann A, Menon S, Raspollini MR, Rubin MA, Srigley JR, Hoon Tan P, Tickoo SK, Tsuzuki T, Turajlic S, Cree I, Moch H. The 2022 World Health Organization Classification of Tumors of the Urinary System and Male Genital Organs-Part B: Prostate and Urinary Tract Tumors. Eur Urol. 2022 Nov;82(5):469-482. doi: 10.1016/j.eururo.2022.07.002. Epub 2022 Aug 11. PMID 35965208